CLINICAL TRIAL: NCT03885882
Title: An Open-Label, Randomized, Single Dose Study to Evaluate the Pharmacokinetics of Three Types of E0302 Sustained Release (SR) Tablets Compared With E0302 Immediate Release (IR) Tablet Under Fed Conditions in Healthy Subjects
Brief Title: A Pharmacokinetic (PK) Study of Three Types of E0302 Sustained Release (SR) Tablets Compared With E0302 Immediate Release (IR) Tablet Under Fed Conditions in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E0302-J064-003
Record Dates: First submitted 2019-03-06; First posted 2019-03-22 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-01

CONDITIONS: Healthy Subjects
Keywords: E0302; Healthy Subjects; E0302 SR Tablet; E0302 IR Tablet

STUDY DESIGN:
Intervention Model Description: Cohort 1 and Cohort 2 will receive treatment as parallel assignment. Cohort 3 will receive treatment in cross-over manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: E0302 Sustained Release (SR1) 1500 mcg (Experimental): Participants will receive a single dose of E0302 SR1 1500 microgram (mcg), tablet, orally on Day 1.
  Interventions: Drug: E0302 SR1
- Cohort 2: E0302 Sustained Release (SR3) 1500 mcg (Experimental): Participants will receive a single dose of E0302 SR3 1500 mcg, tablet on Day 1.
  Interventions: Drug: E0302 SR3
- Cohort 3: E0302 SR2 1500 mcg + E0302 IR 500 mcg (Experimental): Participants will receive a single dose of E0302 SR2 1500 mcg tablet (Treatment A) on Day 1 in Treatment Period 1 followed by single dose of E0302 IR 500 mcg tablet (Treatment B) on Day 7 in Treatment Period 2. A wash-out phase of at least 5 days will be maintained between the treatment periods.
  Interventions: Drug: E0302 SR2; Drug: E0302 IR
- Cohort 3: E0302 IR 500 mcg + E0302 SR2 500 mcg (Experimental): Participants will receive a single dose of E0302 IR 500 mcg tablet (Treatment B) on Day 1 in Treatment Period 1 followed by single dose of E0302 SR2 1500 mcg tablet (Treatment A) on Day 7 in Treatment Period 2. A wash-out phase of at least 5 days will be maintained between the treatment periods.
  Interventions: Drug: E0302 SR2; Drug: E0302 IR

INTERVENTIONS:
Drug: E0302 SR1 — E0302 SR1, oral tablet.
  Arms: Cohort 1: E0302 Sustained Release (SR1) 1500 mcg
Drug: E0302 SR3 — E0302 SR3, oral tablet.
  Arms: Cohort 2: E0302 Sustained Release (SR3) 1500 mcg
Drug: E0302 SR2 — E0302 SR2, oral tablet.
  Arms: Cohort 3: E0302 IR 500 mcg + E0302 SR2 500 mcg; Cohort 3: E0302 SR2 1500 mcg + E0302 IR 500 mcg
Drug: E0302 IR — E0302 IR, oral tablet.
  Arms: Cohort 3: E0302 IR 500 mcg + E0302 SR2 500 mcg; Cohort 3: E0302 SR2 1500 mcg + E0302 IR 500 mcg

SUMMARY:
To assess the PK and safety after administration of three types of E0302 SR tablets (SR1, SR2, SR3) and E0302 IR tablet.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

1. Body mass index (BMI) of 18 to 30 kilogram per meter square [kg/m2], inclusive at Screening

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug test or breath alcohol test at Screening or Baseline
2. Subjects who contravene the restrictions on concomitant medications, food and beverages
3. Currently enrolled in another clinical study or used any investigational drug or device within 3 months preceding informed consent

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for E0302 SR1, SR2, SR3 and IR | Cohort 1 and 2 Day 1: 0-72 hours post dose; Cohort 3 Day 1 or 7: 0-72 hours post dose
AUC (0-t): Area Under the Concentration-Time Curve From Zero Time to Time of Last Quantifiable Concentration | Cohort 1 and 2 Day 1: 0-72 hours post dose, Cohort 3 Day 1 or 7: 0-72 hours post dose
AUC (0 - infinity): Area Under the Concentration-Time Curve From Zero Time Extrapolated to Infinite Time | Cohort 1 and 2 Day 1: 0-72 hours post dose, Cohort 3 Day 1 or 7: 0-72 hours post dose
Number of Participants With Serious Adverse Events (SAEs) and Non-Serious Adverse Events (Non-SAEs) | Cohort 1 and Cohort 2: Up to 12 days, Cohort 3: Up to 18 days
Number of Participants With Abnormal Clinical Laboratory Values | Cohort 1 and Cohort 2: Up to Day 4, Cohort 3: Up to Day 10
Number of Participants With Abnormal Vital Sign Values | Cohort 1 and Cohort 2: Up to Day 2, Cohort 3: Up to Day 8
Number of Participants With Abnormal 12-lead Electrocardiogram Values | Cohort 1 and Cohort 2: Up to Day 12, Cohort 3: Up to Day 18

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland Clinical Studies, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.